CLINICAL TRIAL: NCT02044250
Title: Comparison of Clopidogrel vs. Aspirin Monotherapy Beyond Two Year After Drug-eluting Stent Implantation
Brief Title: Harmonizing Optimal Strategy for Treatment of Coronary Artery Stenosis- EXtended Antiplatelet Monotherapy (HOST-EXAM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical (Industry); Samjin Pharmaceutical Co., Ltd. (Industry); Daewoong Pharmaceutical Co. LTD. (Industry); Hanmi Pharmaceutical co., ltd. (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Principal investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOST-EXAM Trial
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Coronary Heart Disease
Keywords: Aspirin; Clopidogrel; Antiplatelet monotherapy; Drug-eluting stent
MeSH Terms: conditions — Coronary Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Active Comparator): Antiplatelet monotherapy : Clopidogrel 75mg P.O. daily
  Interventions: Drug: Clopidogrel
- Aspirin (Placebo Comparator): Antiplatelet monotherapy : Aspirin 100~200mg P.O. daily
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75mg 1tab P.O. daily
  Other Names: Copregrel, Plateless, Cloart, Pidogul
  Arms: Clopidogrel
Drug: Aspirin — Aspirin 100~200mg 1~2tab P.O. daily
  Arms: Aspirin

SUMMARY:
Objectives :

To compare the efficacy and safety of clopidogrel monotherapy with aspirin monotherapy in patients who received dual or triple antiplatelet therapy for 1 year (± 6 months) after drug-eluting stent implantation for coronary artery disease

Patient Enrollment :

5530 patients enrolled at 55 centers in Korea

Patient Follow-up :

Clinical follow-up will occur at 1, 12 and 24 months.

Primary Endpoint :

Composite endpoint of MACE and major bleeding

Secondary Endpoint :

Device-oriented composite outcome including TLR (target lesion revascularization), TVR (target vessel revascularization), stent thrombosis, and minor GI (gastrointestinal) complications

DETAILED DESCRIPTION:
The primary purpose of this study is to compare the efficacy and safety of antiplatelet monotherapy with aspirin or clopidogrel for 2 years in patients who have not experienced MACE (major adverse cardiac events) including all-cause death, acute coronary syndrome including non-fatal MI (myocardial infarction), or urgent revascularization under combined antiplatelet therapy for 12 ± 6 months after PCI (percutaneous coronary intervention) with DES (drug-eluting stents). The trial tests the hypothesis that clopidogrel is superior to aspirin in preventing clinical events and device-oriented outcomes. Clinical events are defined as a composite of all-cause death, non-fatal MI, stroke, readmission due to acute coronary syndrome (ACS), or Bleeding Academic Research Consortium (BARC) class ≥ 3.29 Device-oriented outcomes include target lesion/vessel revascularization (TLR/TVR) and Academic Research Consortium (ARC)-defined stent thrombosis.

The primary endpoint of this study is the rate of clinical events defined as a composite of MACE and major bleeding complications. MACE includes all-cause death, non-fatal MI, stroke, and readmission due to ACS (acute coronary syndrome). Major bleeding is defined as bleeding (BARC class ≥ 3) at 24 months. Non-fatal MI is defined as any confirmed evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia without resulting in death, which is supported by electrocardiography, cardiac enzymes, or cardiac imaging according to the third Universal Definition of MI.37, 38 A readmission due to ACS is defined as any re-hospitalization definitely originating from an ACS event, which satisfies the definition of the American College of Cardiology Foundation and the American Heart Association.37, 39 A stroke is defined as any abrupt-onset, non-convulsive, focal, or global neurological deficit lasting more than 24 hours, which is caused by ischemia or hemorrhage in the brain.39 Secondary endpoints are the rate of device-oriented outcomes including TLR/TVR and stent thrombosis at 24 months, and minor gastrointestinal (GI) complications with the related cost-effectiveness. TLR is defined as any repeat revascularization procedure at the original lesion of the index procedure any time during the follow-up period.40 TVR is defined as any repeat revascularization procedure involving at least one of the target vessels that were treated in the index procedure.40 Stent thrombosis is defined according to the ARC.41, 42 Minor GI complications are assessed on the basis of newly developed GI symptoms, newly added GI medications, or symptom-driven GI endoscopy. At each visit, clinicians will question the patient regarding GI symptoms from intermittent epigastric soreness or bloating due to melena/hematochezia. Any additional GI medications, including H2-blockers and proton pump inhibitors, will be documented for each patient. If a patient undergoes endoscopy, the type of endoscopy, test results, and further interventions will be recorded. Additional medical costs related to these minor GI complications (South Korean won/year) will be calculated to assess the cost effectiveness of each drug based on average Korean expenses. All endpoints will be assessed primarily by the investigator and adjudicated secondarily by the independent clinical event committee.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged ≥20 years
2. Maintenance of dual or triple antiplatelet therapy at least 12 ± 6 months after PCI with DES
3. No history of further clinical event after PCI with DES
4. Plan to change to antiplatelet monotherapy
5. Agreement to give written informed consent

Exclusion Criteria:

1. History of hypersensitivity to aspirin or clopidogrel
2. History of contraindication to aspirin or clopidogrel
3. Active pathologic bleeding, such as peptic ulcer, tumor bleeding or intracranial hemorrhage
4. History of major bleeding, BARC class ≥3, resulting in stop of antiplatelet agents within 3 months
5. Bleeding diathesis
6. Known coagulopathy or refusal of blood transfusion
7. Presence of non-cardiac comorbidity with life expectancy <2 years from randomization
8. Plan to surgery or intervention which needs to stop antiplatelet agents ≥3 months
9. Females with childbearing potential or breast-feeding
10. Conditions that may result in protocol non-compliance by the committees
11. Co-administration of contraindicated medications as follows: other P2Y 12 inhibitors (prasugrel or ticagrelor); anticoagulants (warfarin, new oral anticoagulants, or chronic therapy of heparin); cytochrome P450 2C19 inhibitors (fluoxetine, moclobemid or voriconazole); probenecid; high dose of methotrexate (≥15 mg/week); lithium
12. Refusal to give written informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5530 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Composite of major adverse cardiovascular events (MACE) and major bleeding complications | 2 years
  MACE, composite of all-cause death, non-fatal MI, stroke, and readmission due to ACS; major bleeding, bleeding of BARC class ≥3

SECONDARY OUTCOMES:
Target vessel revascularization (TVR), target lesion revascularization (TLR) | 2 years
  TVR, any repeat revascularization procedure involving at least one of the target vessels that were treated in the index procedure; TLR, any repeat revascularization procedure at the original lesion of the index procedure
Stent thrombosis (acute, sub-acute, late, very late) | 2 years
  defined according to the ARC
Minor gastrointestinal (GI) complications | 2 years
  newly developed GI symptoms, newly added GI medications, or symptom-driven GI endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Song JE, Yang HM, Kang J, Hwang D, Han JK, Park KW, Kang HJ, Koo BK, Kim HS. Long-term Clopidogrel vs Aspirin Monotherapy in Coronary Artery Disease Patients With High Ischemic Risk: HOST-EXAM Extended Study Post hoc Analysis. Can J Cardiol. 2025 Dec 24:S0828-282X(25)01576-4. doi: 10.1016/j.cjca.2025.11.051. Online ahead of print. PMID 41453443
- [Derived] Han M, Kang J, Kim B, Hwang D, Yang HM, Park KW, Won KB, Han JK, Koo BK, Shin ES, Kim HS. The impact of body mass index on antiplatelet monotherapy strategy for secondary prevention after percutaneous coronary intervention: A substudy of the HOST-EXAM trial. Am Heart J. 2025 Dec;290:258-267. doi: 10.1016/j.ahj.2025.07.005. Epub 2025 Jul 5. PMID 40623657
- [Derived] Kang J, Chung J, Park KW, Bae JW, Lee H, Hwang D, Yang HM, Han KR, Moon KW, Kim U, Rhee MY, Kim DI, Kim SY, Lee SY, Lee SU, Kim SW, Kim SY, Han JK, Shin ES, Koo BK, Kim HS. Long-Term Aspirin vs Clopidogrel After Coronary Stenting by Bleeding Risk and Procedural Complexity. JAMA Cardiol. 2025 May 1;10(5):427-436. doi: 10.1001/jamacardio.2024.4030. PMID 39602157
- [Derived] Yang S, Kang J, Park KW, Hur SH, Lee NH, Hwang D, Yang HM, Ahn HS, Cha KS, Jo SH, Ryu JK, Suh IW, Choi HH, Woo SI, Han JK, Shin ES, Koo BK, Kim HS. Comparison of Antiplatelet Monotherapies After Percutaneous Coronary Intervention According to Clinical, Ischemic, and Bleeding Risks. J Am Coll Cardiol. 2023 Oct 17;82(16):1565-1578. doi: 10.1016/j.jacc.2023.07.031. PMID 37821166
- [Derived] Lee K, Kang J, Park KW, Park TH, Kim BS, Lim SW, Cho YH, Jeon DW, Kim SH, Yang HM, Kang HJ, Han JK, Shin ES, Koo BK, Kim HS. Impact of Age on Antiplatelet Monotherapy in the Chronic Maintenance Period After Percutaneous Coronary Intervention: A Post Hoc Analysis From the HOST-EXAM Extended Study. Can J Cardiol. 2024 Jan;40(1):43-52. doi: 10.1016/j.cjca.2023.09.021. Epub 2023 Sep 22. PMID 37742741
- [Derived] Hwang D, Kim HL, Koo BK, Rhee TM, Yang DW, Seo Y, Byun J, Kang J, Han JK, Park KW, Shin ES, Rha SW, Bae JW, Mamas MA, Cohen DJ, Lee TJ, Kim HS; HOST-EXAM Investigators. Cost-Effectiveness of Clopidogrel vs Aspirin Monotherapy After Percutaneous Coronary Intervention: Results From the HOST-EXAM Study. JACC Asia. 2023 Mar 14;3(2):198-207. doi: 10.1016/j.jacasi.2022.12.007. eCollection 2023 Apr. PMID 37181388
- [Derived] Rhee TM, Bae JW, Park KW, Rha SW, Kang J, Lee H, Yang HM, Kwak SH, Chae IH, Shin WY, Kim DK, Oh JH, Jeong MH, Kim YH, Lee NH, Hur SH, Yoon J, Han JK, Shin ES, Koo BK, Kim HS; HOST-EXAM Investigators. Aspirin vs Clopidogrel for Long-term Maintenance After Coronary Stenting in Patients With Diabetes: A Post Hoc Analysis of the HOST-EXAM Trial. JAMA Cardiol. 2023 Jun 1;8(6):535-544. doi: 10.1001/jamacardio.2023.0592. PMID 37043192
- [Derived] Shin ES, Jun EJ, Kim B, Won KB, Koo BK, Kang J, Park KW, Rhee TM, Yang HM, Han JK, Kim HS; HOST-EXAM Investigators. Association of Clinical Outcomes With Sex in Patients Receiving Chronic Maintenance Antiplatelet Monotherapy After Percutaneous Coronary Intervention: A Post Hoc Gender Analysis of the HOST-EXAM Study. J Am Heart Assoc. 2023 Apr 18;12(8):e026770. doi: 10.1161/JAHA.122.026770. Epub 2023 Apr 12. PMID 37042284
- [Derived] Kang J, Park KW, Lee H, Hwang D, Yang HM, Rha SW, Bae JW, Lee NH, Hur SH, Han JK, Shin ES, Koo BK, Kim HS. Aspirin Versus Clopidogrel for Long-Term Maintenance Monotherapy After Percutaneous Coronary Intervention: The HOST-EXAM Extended Study. Circulation. 2023 Jan 10;147(2):108-117. doi: 10.1161/CIRCULATIONAHA.122.062770. Epub 2022 Nov 7. PMID 36342475
- [Derived] Koo BK, Kang J, Park KW, Rhee TM, Yang HM, Won KB, Rha SW, Bae JW, Lee NH, Hur SH, Yoon J, Park TH, Kim BS, Lim SW, Cho YH, Jeon DW, Kim SH, Han JK, Shin ES, Kim HS; HOST-EXAM investigators. Aspirin versus clopidogrel for chronic maintenance monotherapy after percutaneous coronary intervention (HOST-EXAM): an investigator-initiated, prospective, randomised, open-label, multicentre trial. Lancet. 2021 Jun 26;397(10293):2487-2496. doi: 10.1016/S0140-6736(21)01063-1. Epub 2021 May 16. PMID 34010616